CLINICAL TRIAL: NCT06082986
Title: A Multicenter, Retrospective, Observational Study Using Real-world Data to Describe the Effectiveness, Treatment Pattern and Safety of Ustekinumab Among Bio-naive Patients With Crohn's Disease in China
Brief Title: A Retrospective Observational Study of Ustekinumab Among Bio-naive Participants With Crohn's Disease in China
Status: Completed | Type: Observational
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR109344; PCSIMMA0055 (Other: Xian-Janssen Pharmaceutical Ltd., China)
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bio-naive Participants With Crohn's Disease (CD): Participants with CD from inflammatory bowel disease (IBD) database who received ustekinumab from 20 May 2020 to 16 September 2022 in the real-world setting in China will be observed in the study. Only data available per routine clinical practice will be collected within this study.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — No interventions will be administered as a part of this study. Participants received ustekinumab as per their routine clinical practice.

SUMMARY:
Bio-naive participants are defined as the participants who previously have not received any biologics for Crohn's Disease (CD).The purpose of this retrospective study is to describe the endoscopic remission at week 24 among bio-naive participants with CD treated with ustekinumab in China.

ELIGIBILITY:
Inclusion Criteria:

* Participants with diagnosis of active Crohn's Disease (CD) (that is, Crohn's Disease Activity Index [CDAI] greater than or equal to [>=] 150; Harvey-Bradshaw Index [HBI] >=5; or determined by physicians)
* Participants with initiation of ustekinumab intravenous induction therapy for the first time between 20 May 2020 and 16 September 2022

Exclusion Criteria:

* Previously received ustekinumab for any indication other than CD
* Participants were previously exposed with any biologics (for example: adalimumab, infliximab, vedolizumab or their biosimilars) other than ustekinumab

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population will consist of bio-naive participants who initiated ustekinumab therapy for the first time between 20 May 2020 and 16 September 2022.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Endoscopic Remission at Week 24 | Week 24
  Endoscopic remission: simple endoscopic score for crohn's disease (SES-CD) less than or equal to (<=) 2, total SES-CD <=4, a decrease in total SES-CD greater than or equal to (>=) 2 from baseline, and no subtotal SES-CD >1 for each endoscopic parameter (for isolated ileal, ileocolonic and isolated colonic CD), rutgeerts score <=i1 (for post-operation CD). SES-CD: assesses disease severity based on 4 endoscopic parameters across 5 ileocolonic segments. Total SES-CD = 0 to 56,higher scores = more severe disease. Rutgeerts score: assess postoperative disease recurrence with no lesions (i0); <=5 aphthous lesions (i1); >5 aphthous ulcers with normal intervening mucosa/patchy areas of larger lesions/lesions confined to ileocolic anastomosis (i2); diffuse aphthous ileitis and diffusely inflamed mucosa (i3); diffuse inflammation with large ulcers, nodules, and/or stenosis (i4).

SECONDARY OUTCOMES:
Percentage of Participants With Endoscopic Response at Week 24 | Week 24
  Endoscopic response is defined as >50 percent (%) decrease from baseline in total SES-CD. The SES-CD is a scoring system to assess disease severity in participants with CD. The SES-CD score is based on the evaluation of 4 endoscopic components: size of ulcers, surface ulceration, affected surface size, and presence of luminal narrowing across 5 predefined ileocolonic segments (ileum, right colon, transverse colon, left colon and rectum). Each component score= 0 to 3 for each segment with total SES-CD score ranges from 0 to 56, where higher scores indicates more severe disease.
Percentage of Participants With Clinical Remission at Week 24 | Week 24
  Clinical remission is achieved when total crohn's disease activity index (CDAI) <150 or total of harvey-bradshaw index (HBI) score <5. CDAI assesses CD based on variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain, use of antidiarrheal drug(s) and general well-being. CDAI score: asymptomatic remission: <150, mild: 150-220, moderate: 221-450, severe: >450. HBI parameters: general well-being (0-4, higher score means lower well-being), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day (score 1 per movement), abdominal mass (0=none, 1=dubious, 2=definite, 3=definite and tender) and complications (score 1 per item). Total score is sum of individual parameters. Score ranges from 0 to no pre-specified maximum score as it depends on number of complications and liquid stools per day. HBI score: <5 (remission), 5-7 (mild disease), 8-16 (moderate disease) and >16 (severe disease).
Percentage of Participants With Clinical Response at Week 24 | Week 24
  Clinical response is defined as decrease in total CDAI score from >=100 or a CDAI score <150 or decrease in total HBI score >=3 from baseline. CDAI assesses CD based on variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain, use of antidiarrheal drug(s) and general well-being. CDAI score: asymptomatic remission: <150, mild: 150-220, moderate: 221-450, severe: >450. HBI parameters: general well-being (0-4, higher score means lower well-being), abdominal pain (0-3, higher score=more severe pain), number of liquid stools per day (score 1 per movement), abdominal mass (0=none, 1=dubious, 2=definite, 3=definite and tender) and complications (score 1 per item). Total score is sum of individual parameters. Score ranges from 0 to no pre-specified maximum score as it depends on number of complications and liquid stools per day. HBI score: <5 (remission), 5-7 (mild disease), 8-16 (moderate disease) and >16 (severe disease).
Percentage of Participants With Steroid-free Clinical Remission at Week 24 | Week 24
  Steroid-free clinical remission is achieved when total CDAI score <150 or total HBI score <5, without use of any steroid preparations. CDAI assesses CD based on variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain, use of antidiarrheal drug(s) and general well-being. CDAI score: asymptomatic remission: <150, mild: 150-220, moderate: 221-450, severe: >450. HBI parameters: general well-being (0-4, higher score=lower well-being), abdominal pain (0-3, higher score=more severe pain), number of liquid stools per day (score 1 per movement), abdominal mass (0=none, 1=dubious, 2=definite, 3=definite and tender) and complications (score 1 per item). Total score is sum of individual parameters. Score ranges from 0 to no pre-specified maximum score as it depends on the number of liquid stools per day and number of complications. HBI score: <5 (remission), 5-7 (mild disease), 8-16 (moderate disease) and >16 (severe disease).
Percentage of Participants With Steroid-free Clinical Response at Week 24 | Week 24
  Steroid-free clinical response: decrease in total CDAI score >=100 or total HBI score >=3 from baseline, without use of any steroid preparations. CDAI assesses CD based on variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain, use of antidiarrheal drug(s) and general well-being. CDAI score: asymptomatic remission: <150, mild: 150-220, moderate: 221-450, severe: >450. HBI parameters: general well-being (0-4, higher score=lower well-being), abdominal pain (0-3, higher score=more severe pain), number of liquid stools per day (score 1 per movement), abdominal mass (0=none, 1=dubious, 2=definite, 3=definite and tender) and complications (score 1 per item). Total score is sum of individual parameters. Score ranges from 0 to no pre-specified maximum score as it depends on number of complications and liquid stools per day. HBI score: <5 (remission), 5-7 (mild disease), 8-16 (moderate disease) and >16 (severe disease).
Change From Baseline in C-Reactive Protein (CRP) at Week 24 | Baseline and Week 24
  Change from baseline in CRP at Week 24 will be reported.
Change From Baseline in Fecal Calprotectin at Week 24 | Baseline and Week 24
  Change from baseline in fecal calprotectin at Week 24 will be reported.
Percentage of Participants With Disease Progression | From index date up to death or end of study (up to 34.4 months)
  Disease progression is defined as the first occurrence of CD complications, or CD-related surgery and hospitalization from index date to death or end of study. Index date is defined as the date of initiating ustekinumab treatment for the first time. CD-related surgery is defined as the first occurrence of any CD-related intestinal and perianal procedures. CD-related hospitalization is defined as the first occurrence of any CD-related admission, with causes including disease relapse, complication, and drug side effects, except for CD-related surgery.
Time to Disease Progression | From index date up to death or end of study (up to 34.4 months)
  Disease progression is defined as the first occurrence of CD complications, or CD-related surgery and hospitalization from index date to death or end of study. Index date is defined as the date of initiating ustekinumab treatment for the first time. CD-related surgery is defined as the first occurrence of any CD-related intestinal and perianal procedures. CD-related hospitalization is defined as the first occurrence of any CD-related admission, with causes including disease relapse, complication, and drug side effects, except for CD-related surgery.
Percentage of Participants With Ustekinumab Therapy Switch During the Observational Period to Other Therapy | From index date up to death or end of study (up to 34.4 months)
  Percentage of participants who will switch to other therapy will be reported. Therapy switch is defined as switching to other biologic therapy from index date to death or end of study. Index date is defined as the date of initiating ustekinumab treatment for the first time.
Percentage of Participants With Reasons for Ustekinumab Therapy Switch to Other Therapy | From index date up to death or end of study (up to 34.4 months)
  Percentage of participants with reasons for ustekinumab therapy switch to other therapy will be reported. Therapy switch is defined as switching to other biologic treatments from index date to death or end of study. Index date is defined as the date of initiating ustekinumab treatment for the first time.
Percentage of Participants With Ustekinumab Therapy Discontinuation | From index date up to death or end of study (up to 34.4 months)
  Percentage of participants with ustekinumab therapy discontinuation will be reported. Therapy discontinuation is defined as having a ustekinumab therapy gap of greater than or equal to (>=) 120 days without treatment switch or intravenous re-induction from index date to death or end of study. Index date is defined as the date of initiating ustekinumab treatment for the first time.
Percentage of Participants With Reasons for Ustekinumab Therapy Discontinuation | From index date up to death or end of study (up to 34.4 months)
  Percentage of participants with reasons for ustekinumab therapy discontinuation will be reported. Therapy discontinuation is defined as having a ustekinumab therapy gap of >=120 days without treatment switch or intravenous re-induction from index date to death or end of study. Index date is defined as the date of initiating ustekinumab treatment for the first time.
Time to Ustekinumab Therapy Switch or Discontinuation | From index date up to death or end of study (up to 34.4 months)
  Time to ustekinumab therapy switch or discontinuation will be reported. Therapy switch is defined as switching to other biologic therapy from index date to death or end of study. Therapy discontinuation is defined as having a ustekinumab therapy gap of >=120 days without treatment switch or intravenous re-induction from index date to death or end of study. The time to therapy switch or discontinuation is defined as follows: 1) For participants with an event date, it is calculated as the difference between the event date and index date, adding 1. 2) For participants without an event date, it is calculated as the difference between the end of the observation date (death/end of study) and the index date, adding 1; this time is a censoring time. The event date is the initiation date of therapy switch or discontinuation, whichever happens first. Index date is defined as the date of initiating ustekinumab treatment for the first time.
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From index date up to death or end of study (up to 34.4 months)
  Percentage of participants with AEs and SAEs will be reported. An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Index date is defined as the date of initiating ustekinumab treatment for the first time.
Percentage of Participants With Each Adverse Event (AE) | From index date up to death or end of study (up to 34.4 months)
  Percentage of participants with each AE will be reported. An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. Index date is defined as the date of initiating ustekinumab treatment for the first time.
Duration of Each Adverse Event (AE) | From index date up to death or end of study (up to 34.4 months)
  Duration of each AE will be reported. Duration of each AE's is defined as time from onset of AE to end date of each AE or till the end of the study. An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. Index date is defined as the date of initiating ustekinumab treatment for the first time.
Percentage of Participants With Each AE's Outcome | From index date up to death or end of study (up to 34.4 months)
  Percentage of participants with each AE's outcome will be reported. Each AE's outcome includes recovered/resolved, recovered/resolved with sequelae, recovering/resolving, not recovered/not resolved, fatal, and unknown. An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. Index date is defined as the date of initiating ustekinumab treatment for the first time.
Percentage of Participants With Ustekinumab Therapy Switch or Discontinuation due to AEs | From index date up to death or end of study (up to 34.4 months)
  Percentage of participants with ustekinumab therapy switch or discontinuation due to AEs will be reported. Therapy switch is defined as switching to other biologic therapy from index date to death or end of study. Therapy discontinuation is defined as having a ustekinumab therapy gap of >=120 days without treatment switch or intravenous re-induction from index date to death or end of study. Index date is defined as the date of initiating ustekinumab treatment for the first time. An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (3):
- China (3):
  - Sir Run Run Shaw Hospital, affiliated with Zhejiang University, School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou

IPD SHARING:
Plan to Share IPD: No